CLINICAL TRIAL: NCT00140491
Title: Visual Field Defects in Non-Arteritic Anterior Ischemic Optic Neuropathy: Effect of Vision Restoration Therapy (VRT)
Brief Title: Vision Restoration Therapy (VRT) to Treat Non-Arteritic Anterior Ischemic Optic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Valerie Biousse, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0435-2005; Valerie Biousse 404-778-5158
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Non-Arteritic Anterior Ischemic Optic Neuropathy
Keywords: Non-Arteritic Anterior Ischemic Optic Neuropathy; Visual Field Defect; Neuroplasticity; Rehabilitation

INTERVENTIONS:
Device: Vision Restoration Therapy (NOVAVISION)

SUMMARY:
The goal of this pilot study is to evaluate the effect of Vision Restoration Therapy, VRT, on the visual function of patients with unilateral or bilateral AION, who have good central vision (at least 20/60) and altitudinal visual field defects.

DETAILED DESCRIPTION:
Anterior ischemic optic neuropathy (AION) is one of the most common causes of optic neuropathy after the age of 50. There is currently no available treatment and although up to 40% of patients have some spontaneous improvement within the first few months, most patients remain visually devastated. About 50% of patients retain relatively spared central visual acuity with an inferior altitudinal visual field defect. These patients usually complain of difficulty reading and loss of depth perception.

Recently, training-induced enlargement of visual field defects has been demonstrated in some patients with VF defects secondary to lesions of the retrochiasmal visual pathways. This computer-based Vision Restoration Therapy (VRT) was developed in Germany and has been FDA-cleared in the United States for the past one year.

VRT is currently available at Emory for patients with homonymous hemianopia. Patients work on personally-designed software (on a laptop at home) twice daily (30 minutes each) for 6 months. Zones of partially damaged neurons, which are usually located between the intact and damaged area of the visual field (transition zone) are deliberately stimulated by VRT. There is only anecdotal evidence that this visual restoration therapy may be helpful in enlarging the visual field of patients with optic neuropathies.

The goal of this pilot study is to evaluate the effect of VRT on the visual function of patients with unilateral or bilateral AION, who have good central vision (at least 20/60) and altitudinal visual field defects. The effect of VRT will be evaluated by visual acuity, color vision, stereo vision, Humphrey VF (24-2 SITA standard) testing, and scales evaluating reading speed and vision-based quality of life. These measures will be repeated before VRT, at 3 months, at 6 months, and at 1 year after VRT. 20 patients will be included in the study. Patients will be randomized at inclusion between VRT and sham (placebo)-training (10 in each group). The 10 patients receiving sham training will then receive VRT for the following 6 months if they so choose. All data will be analyzed in a blinded fashion. The company developing VRT in the United States (NOVAVISION) has agreed to provide VRT and sham-training.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by Dr Biousse or Dr Newman in the Neuro-Ophthalmology Unit at Emory University.
* Age ≥ 30 years.
* Diagnosis of non-arteritic ischemic optic neuropathy at least 6 months prior to inclusion.
* Uni- or bilateral AION (in case of bilateral AION, only one eye will be included in the study).
* Best corrected visual acuity of at least 20/60 in the study eye
* Altitudinal or arcuate visual field defect, splitting fixation by >10 decibel difference above and below horizontal meridian.
* Stable visual function demonstrated by more than two stable visual acuity measurements and two automated visual field testings prior to inclusion in the study.
* Patient willing, and able, to spend 60 minutes-a-day for 6 months working on a computer.

Exclusion Criteria:

* Patient cognitively or physically unable to perform reliable automated perimetry testing (on the 24-2 SITA Standard program) (which is grossly equivalent to the effort and attention needed to perform VRT daily at home).
* Other cause of optic neuropathy.
* Associated ocular disease requiring treatments or responsible for visual loss (such as untreated significant cataract, glaucoma, age related macular degeneration, etc…).
* Visual acuity worse than 20/60 in the study eye.
* Non-stable visual field defect on previous evaluations.
* Epilepsy.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Visual Function

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Biousse, MD, Principal Investigator — Emory Eye Center
Locations (1):
- Emory Eye Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Jung CS, Bruce B, Newman NJ, Biousse V. Visual function in anterior ischemic optic neuropathy: effect of Vision Restoration Therapy--a pilot study. J Neurol Sci. 2008 May 15;268(1-2):145-9. doi: 10.1016/j.jns.2007.12.001. Epub 2008 Jan 22. PMID 18207164